CLINICAL TRIAL: NCT00876798
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of Oral Lixivaptan Capsules in Subjects With Euvolemic Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CardioKine Inc. (Industry)
Collaborators: Cardiokine Biopharma, LLC (Industry); Biogen (Industry)
Responsible Party: Cesare Orlandi, MD, Cardiokine Biopharma LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CK-LX3430
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-11

CONDITIONS: Euvolemic Hyponatremia
Keywords: Euvolemic Hyponatremia; SIADH; Serum Sodium
MeSH Terms: conditions — Inappropriate ADH Syndrome | interventions — lixivaptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lixivaptan
  Interventions: Drug: Lixivaptan
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lixivaptan — Capsules, 25mg lixivaptan or matching placebo once daily. Study medication can be titrated up to 50mg or 100mg once daily. Acceptable dosages are once daily administration of 25mg, 50mg, or 100mg as a single dose.
  Arms: 1
Drug: Placebo — Capsule. Subjects will be randomized (3:1) on an outpatient basis to 25 mg lixivaptan or matching placebo, once daily.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of oral lixivaptan capsules in subjects with Euvolemic Hyponatremia.

DETAILED DESCRIPTION:
Phase I and Phase II clinical trials have demonstrated that lixivaptan may play an important role in treating hyponatremia and the signs and symptoms of water retention associated with HF, LCWA, and SIADH. Lixivaptan was previously evaluated in disease states characterized by hyponatremia with euvolemia (SIADH) and hyponatremia combined with fluid overload (HF, LCWA). Lixivaptan demonstrated correction in serum sodium concentration together with marked aquaresis in subjects with hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Men or women aged 18 or older.
3. Diagnosis of euvolemic hyponatremia (Na+ < 135 mEq/L).
4. Willing to be observed in a monitored setting for approximately the first 8 hours following treatment initiation (first dose).
5. In the Investigator's judgement the patient has adequate visual and auditory acuity to allow participation in the trial.

Exclusion Criteria:

1. Pregnant or breast-feeding women, or women planning to become pregnant or to breastfeed.
2. Overt symptoms of hyponatremia requiring immediate medical intervention (e.g., coma, seizures).
3. Acute or transient hyponatremia (e.g., associated with head trauma, postoperative state, or use of radiotherapy and/or chemotherapy).
4. Hyponatremia in hypovolemic states (e.g., due to fluid loss through vomiting, diarrhea, burns, etc.). Hypovolemic hyponatremia is defined as the presence of clinical evidence of extracellular fluid volume depletion.
5. Hyponatremia in hypervolemic states (e.g., congestive heart failure). Hypervolemia is defined as a presence of increased total body water with signs of edema.
6. Pseudohyponatremia (i.e., hyponatremia resulting from a laboratory artifact).
7. Hypertonic hyponatremia (e.g., hyponatremia in the setting of hyperglycemia).
8. Hyponatremia as a result of any medication that can safely be withdrawn.
9. Hyponatremia due to hypothyroidism or adrenal insufficiency.
10. Current diagnosis of psychogenic polydipsia.
11. Receiving within 7 days of enrollment other medication for treatment of hyponatremia, specifically: demeclocycline, lithium carbonate, urea, or any vasopressin antagonist.
12. Supine systolic arterial blood pressure of ≤ 90 millimeters of mercury (mmHg).
13. Serum creatinine > 3.0 mg/dL (> 265.2 mol/L).
14. Hypokalemia based on clinical sign/symptoms or lab findings (e.g., serum potassium < 3.5 mEq/L).
15. Uncontrolled diabetes mellitus as defined by the Investigators (e.g., hemoglobin - glycosylated [HbA1c] > 9%).
16. ST-segment elevation myocardial infarction (STEMI) within 30 days or active myocardial ischemia at the time of enrollment.
17. History of cerebral vascular accident (CVA) within 30 days prior to screening.
18. Severe malnutrition in the Investigator's judgment (e.g., body mass index [BMI] < 17).
19. Advanced liver disease or documented diagnosis of cirrhosis or alcoholic hepatitis.
20. Urinary tract obstruction (benign prostatic hypertrophy [BPH] allowed if non-obstructive).
21. History of chronic drug/medication abuse within the past 6 months or current alcohol abuse.
22. Terminally ill or moribund condition with little chance of short-term survival.
23. Receiving vasopressin or its analogs for treatment of any condition.
24. Known allergy to any vasopressin antagonist.
25. Previous participation in a lixivaptan study.
26. Recipient of any investigational treatment within 30 days prior to baseline visit.
27. Unable to take oral medications.
28. Significant neurological disorders (e.g., permanent neurological deficits, probable Alzheimer's disease, normal pressure hydrocephalus, Parkinsonian dementia complex, multi-infarct dementia, mixed dementia, or Huntington's disease).
29. Conditions limiting access to water or an inability to respond to thirst (e.g., hydrophobia, or non-communicative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To demonstrate that lixivaptan is safe and effective in achieving and maintaining increased serum sodium concentration in subjects with SIADH and other conditions of euvolemic hyponatremia. | 6 months

SECONDARY OUTCOMES:
If lixivaptan demonstrates improvement in serum sodium, % of subjects achieving normalized serum sodium, % of subjects requiring fluid restriction, prevention of worsening hyponatremia, and the change from baseline to complete TMT-B. | 6 months

CONTACTS AND LOCATIONS:
Locations (90):
- United States (66):
  - Birmingham Nursing and Rehabilitation East, Birmingham, Alabama
  - Healthscan Research, LLC, Montgomery, Alabama
  - PsyPharma Clinical Research, Inc., Phoenix, Arizona
  - PsyPharma Clinical Research, Phoenix, Arizona
  - Southern Arizona VA Health Care System (SAVAHCS), Tucson, Arizona
  - Parkview Rehabilitation and Nursing, Little Rock, Arkansas
  - Searcy Medical Center, Searcy, Arkansas
  - AV Institute, Inc., Carson, California
  - Royal Care Nursing Home, Fountain Valley, California
  - Sarah S. Olelewe, MD, Inc., Hawthorne, California
  - Torrance Clinical Research, Lomita, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Senior Care of Colorado, PC, Aurora, Colorado
  - Naples Institute for Clinical Research, Bonita Springs, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Jacksonville Center for CLinical Research, Jacksonville, Florida
  - Miami Jewish Home and Hospital for the Aged, Miami, Florida
  - Galiz Research, Miami, Florida
  - Nephrology Associates of South Miami, Miami, Florida
  - Galiz Research, Miami Springs, Florida
  - Piedmont Clinical Trials, North Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Universal Clinical Research & Technology, Inc., Orlando, Florida
  - University Clinical Research & Technology, Inc., Orlando, Florida
  - Coastal Nephrology Associates Reserach Center, Port Charlotte, Florida
  - Executive Health and Research Associates, Atlanta, Georgia
  - Rockdale Medicall Research Associates, Conyers, Georgia
  - RTR Medical Group, Savannah, Georgia
  - Toulon Health Care Center, Toulon, Illinois
  - Research Integrity, LLC, Owensboro, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Natchitoches Internal Medicine, Natchitoches, Louisiana
  - John J. Hainkel Jr Home and Rehabilitation Center, New Orleans, Louisiana
  - Levindale Hebrew Geriatric Center and Hospital, Baltimore, Maryland
  - LifeBridge Health, Inc./ Courtland Gardens Nursing & Rehabilitation Center, Baltimore, Maryland
  - Stephen R. Smith, Baltimore, Maryland
  - Genesis Clinical Research & Consulting, LLC, Fall River, Massachusetts
  - Western New England Renal & Transplant Assciates, PC, Springfield, Massachusetts
  - Millenium Psychiatric Associates, St Louis, Missouri
  - SLU Care Doctors Office Building, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Internal Medical Associates of Grand Island, PC, Grand Island, Nebraska
  - Buffalo VA Medical Center, Buffalo, New York
  - Erie County Medical Center/SUNY at Buffalo affiliate, Buffalo, New York
  - Parker Jewish Institute for Health Care and Rehabilitation, New Hyde Park, New York
  - Rochester General Hospital, Rochester, New York
  - Medical Research Development Associates, LLC, Springfield Gardens, New York
  - Three Rivers Health and Rehabilitation, Windsor, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Valley Medical Research, Centerville, Ohio
  - Hilltop Physicians Inc, Cincinnati, Ohio
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - COR Clinical Research LLC, Oklahoma City, Oklahoma
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Translational Neuroscience, LLC/Drexel University College of Medicine, Conshohocken, Pennsylvania
  - Ilumina CLinical Associates, Indiana, Pennsylvania
  - Carolina Diabetes and Kidney Center, Sumter, South Carolina
  - Senior Adults Specialty Research, Austin, Texas
  - Memorial Hermann - Memorial City Research Center, Houston, Texas
  - South Texas Institutes of Health, McAllen, Texas
  - InVisions Consultants, LLC, San Antonio, Texas
  - ASpen CLinical Research, Orem, Utah
  - Clinical Research and Consulting Center, Fairfax, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Universal Research Group, Tacoma, Washington
- Hospital Erasme, Bruzelles, Bruzelles, Belgium
- Czechia (2):
  - Fakultni nemocnice Ostrava Neurologicke oddeleni, Ostrava, Poruba
  - Klinika nefrologie VFN a 1.LF UK, Nemocnice 2, Prague
- India (10):
  - Smt G.R. Doshi & Smt K.M. Mehta Institute of Kidney Diseases & Reseacrh Cnetre (IKDRC) & Dr. H.L. Trivedi Institute of Transplantation Services (ITS), Asarwa, Ahmedabad
  - Kamineni Hospitals, Hyderabad, Andhra Pradesh
  - Apollo Hospitals, Tanil Nadu, Chennai
  - Kovai Medical Centre & Hospital, Tamil Nadu, Coimbatore
  - M. S. Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Dayanand Medical College and Hospital, Tagorenagar, Ludhiana
  - Bhatia Hospital, G-1 Ward, Mumbia, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - Justice K. S. Hedge Charitable Hospital, Karnataka, Mangalore
  - Department of Neurology St. John's Medical College & Hospital, Bangalore
- Israel (4):
  - Hadassah Medical Organization, Hadassah University Hospital, Ein Karem, Kiryat Hadassah, Jerusalem
  - Diabetic and Endocrine Unit, Hillel Yaffe Medical Center, Hadera
  - The Endocrine Institute, Rabin Medical Center, Beilinson Hospital, Petah Tikvah
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - Presidio ospedaliero zona aretina, Ospedale San Donato di Arezzo, Pietro Nenni, Arezzo
  - SOD Clinica di Endocrinologia a Malatte del Metabolismo, Torette Di Ancona, Torette Di Ancona
  - Medicina II, Arcispedale Santa Maria Nuova, Reggio Emilia
- Mexico (2):
  - Hospital General "Dr. Santiago Ramon Y Cajal" I.S.S.S.T.E., Durango, Mexico
  - Instituto Biomedico de Investigacion A.C., Aguascalientes
- Peru (2):
  - Hospital Nacional Guillermo Almenara Irigoyen-EsSalud., Lima, Peru
  - Hospital Nacional Arzobispo Loayza, Lima, Peru